CLINICAL TRIAL: NCT07102498
Title: A Comparison of Units Used for Blood Glucose and HbA1c Testing
Brief Title: A Comparison of Different Units for Blood Glucose (mmol/L and mg/dl) and Hemoglobin A1c (% and mmol/Mol) Results.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: units
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- bgmmol a1cpercent (Placebo Comparator): BG presented in mmol/L and HbA1c presented in percent
  Interventions: Behavioral: BG mmol/L; Behavioral: A1c percent
- bgmmol a1cmmol (Experimental): BG presented in mmol/L and HbA1c presented in mmol/mol
  Interventions: Behavioral: BG mmol/L; Behavioral: A1c mmol/mol
- bgmgdl a1cpercent (Experimental): BG presented in mg/dl and HbA1c presented in percent
  Interventions: Behavioral: BG mg/dl; Behavioral: A1c percent
- bgmgdl a1cmmol (Experimental): BG presented in mg/dl and HbA1c presented in mmol/mol
  Interventions: Behavioral: BG mg/dl; Behavioral: A1c mmol/mol

INTERVENTIONS:
Behavioral: BG mmol/L — BG presented in mmol/L (the standard presentation in Canada)
  Arms: bgmmol a1cmmol; bgmmol a1cpercent
Behavioral: BG mg/dl — BG presented in mg/dl
  Arms: bgmgdl a1cmmol; bgmgdl a1cpercent
Behavioral: A1c percent — HbA1c presented in percent (the standard presentation in Canada)
  Arms: bgmgdl a1cpercent; bgmmol a1cpercent
Behavioral: A1c mmol/mol — HbA1c presented in mmol/mol
  Arms: bgmgdl a1cmmol; bgmmol a1cmmol

SUMMARY:
A comparison of people's reactions to hypothetical test results using different units.

DETAILED DESCRIPTION:
Comparing how people respond to hypothetical blood glucose results in mg/dl units versus mmol/L units, and also how they respond to hypothetical HbA1c results in % units versus mmol/mol units.

ELIGIBILITY:
Inclusion Criteria:

* Able to use a computer
* Able to use the internet
* Able to read and respond to questions in English or French
* Adults 18+ years old living in Canada

Exclusion Criteria:

- Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Opinion about result | Immediately after the intervention
  Participants' views about the results presented in different units. The exact question wording is: "In your view and based only on the information you have, what is your opinion of this result?" Participants indicate their response on a visual analog scale (a slider) from 0 to 100 with labels "It is not a problem at all" = 0, "I don't know" = 50, or "It is a big problem" = 100.

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on Borealis.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: IPD and supporting information will be shared as soon as the study report is complete and will be available indefinitely.
Access Criteria: Anyone with internet access will be able to access public-facing data. Some data may be restricted to those who register with Borealis.
URL: https://borealisdata.ca/